CLINICAL TRIAL: NCT00855725
Title: Affective Processing in Depression and Epilepsy; An fMRI Study
Brief Title: Affective Processing in Depression and Epilepsy
Status: Terminated | Type: Observational
Why Stopped: PI wanted to discontinue study.
Sponsor: Northwell Health (Other)
Responsible Party: Alan Ettinger, M.D., Vice Chairman, Department of Neurology
Other Study IDs: GCRC 0246; 08-128
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Epilepsy; Depression; Healthy
Keywords: Epilepsy; Depression; Neurology; fMRI; Healthy Controls
MeSH Terms: conditions — Epilepsy; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: fMRI — Subjects will undergo MRI scanning to gather data about cognetive functions.
Other: Hamilton Depression Rating Scale — Investigator will evalute the subject during a one on one interview for depression using the Hamilton Depression Rating Scale.
Other: Beck's Depressive Inventory — Subjects will complete self assessment to evaluate their level of depression.
Other: Interictal Dysphoric Disorder Inventory (IDDI) — Subject will complete self assessment to determine if there have been any changes in mood, emotions and or feelings from time to time.

SUMMARY:
The goal of this study is to determine whether there are unique markers on neuroimaging that are associated with depression in epilepsy.

DETAILED DESCRIPTION:
Symptoms of depression is commonly seen in patients with epilepsy. There are similarities and differences between depressive symptoms in epilepsy when compared with primary depression. Through the use of fMRI (Functional MRI), we hope to determine whether there are unique markers on neuroimaging that are associated with depression in epilepsy.

ELIGIBILITY:
For Control Group

Inclusion Criteria:

* Healthy adults of 18 years of age or older.

Exclusion Criteria:

* Subject has no history of affective disorders
* Subject scores higher than 5 on Hamilton Depression Rating Scale
* Subject with prior primary diagnosis of any psychotic disorder, bipolar disorder, anxiety disorder, or any other serious medical or neurological disorder
* Subject is pregnant
* Subject is unable to undergo a MRI

Epilepsy Only Group

Inclusion Criteria:

* Subject is at least 18 years of age
* Subject has confirmed temporal lobe epilepsy (TLE)

Exclusion Criteria:

* Subject has a history of depression
* Subject scores higher then 5 on Hamilton Depression Rating Scale
* Subject with prior primary diagnosis of any psychotic disorder, bipolar disorder, anxiety disorder, or any other serious medical or neurological disorder
* Subject is pregnant
* Subject is unable to undergo a MRI

Depression Only Group

Inclusion Criteria:

* Subject is at least 18 years of age
* Subject scores between 12 and 18 on Hamilton Depression Rating Scale

Exclusion Criteria:

* Subject scores higher than 18 on Hamilton Depression Rating Scale
* Subject is currently being medicated for depression
* Subject has history of major depression or dysthymia
* Subject with prior primary diagnosis of any psychotic disorder, bipolar disorder, anxiety disorder, or any other serious medical or neurological disorder
* Subject is pregnant
* Subject is unable to undergo a MRI

Depression and Epilepsy Group

Inclusion Criteria:

* Subject has confirmed temporal lobe epilepsy (TLE)
* Subject scores between 12 and 18 on Hamilton Depression Rating Scale

Exclusion Criteria:

* Subject has history of major depression or dysthymia
* Subject is currently on medication for depression
* Subject with prior primary diagnosis of any psychotic disorder, bipolar disorder, anxiety disorder, or any other serious medical or neurological disorder
* Subject is pregnant
* Subject is unable to undergo a MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are four study groups.
  1. Healthy Controls
  2. Subjects with epilepsy only
  3. Subjects with primary depression only
  4. Subjects with epilepsy and depressive symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ettinger, M.D., Principal Investigator — Northwell Health
Locations (1):
- North Shore LIJ Health System, Manhasset, New York, United States